CLINICAL TRIAL: NCT05637398
Title: Colchicine in Patients With Heart Failure and Preserved Left Ventricular Ejection Fraction
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 03-22
Record Dates: First submitted 2022-11-05; First posted 2022-12-05 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-01

CONDITIONS: HFpEF - Heart Failure With Preserved Ejection Fraction; Colchicine
MeSH Terms: interventions — Colchicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All core-laboratory staff will be blind to the endpoints
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine 0.5 bid (Active Comparator): Eligible HFpEF patients will be randomized in 1:1 ratio by an investigator with either colchicine 0.5 twice daily or usual care for 12 weeks
  Interventions: Drug: Colchicine
- Usual Care (No Intervention): Eligible HFpEF patients will be randomized in 1:1 ratio by an investigator with either colchicine 0.5 twice daily or usual care for 12 weeks

INTERVENTIONS:
Drug: Colchicine — The active treatment intervention consists of colchicine 0.5 mg twice daily that will be administrated by the investigator
  Arms: Colchicine 0.5 bid

SUMMARY:
Heart failure with preserved left ventricular ejection fraction (HFpEF) is a syndrome associated with high morbidity and mortality rates. Systemic low-grade inflammation is acknowledged to be a fundamental pathophysiological mechanism of HFpEF. Interventions targeting inflammatory pathway is understudied in HFpEF. Colchicine is a safe and well tolerated anti-inflammatory drug, which interferes with several steps in the inflammatory process. The drug has been extensively studied in different cardiovascular pathologies except HFpEF. We assume that colchicine decreases inflammation and reduces sST2 levels in HFpEF.

DETAILED DESCRIPTION:
HFpEF is a syndrome associated with high morbidity and mortality rates. The underlying mechanisms of the syndrome are not fully understood. Systemic low-grade inflammation is acknowledged to be a fundamental pathophysiological mechanism of HFpEF, which facilitates cardiomyocyte stiffness and myocardial fibrosis development. However, anti-inflammatory treatment approaches are largely under studied. Colchicine is a safe and well tolerated anti-inflammatory drug, which interferes with several steps in the inflammatory process, resulting in suppression of a number of pro-inflammatory pathways and cytokines release, including IL-1, hsCRP. The drug has been extensively studied in patients with coronary artery disease (COLCOT, LoDoCo2) and showed significant reduction in risk of cardio-vascular events, as well as inflammation. Post-hoc analysis of in the CANTOS study investigated the effect of monoclonal antibody targeting interleukin-1β in patients with prior myocardial infarction, showed a reduction in heart failure (HF) hospitalization of patients with elevations in high-sensitivity C-reactive protein (hsCRP). There is no data available regarding the effect of Colchicine on HFpEF patients. Soluble suppression of tumourigenicity 2 (sST2), a member of the interleukin (IL)-1 receptor family, which is not restricted to inflammation, but is also expressed in cardiomyocytes, fibroblast and endothelial cells of cardiac microvessels in response to myocardial stress antagonizing cardioprotective effects of IL-33/ST2 system. In HFpEF, sST2 associated with worse clinical signs and symptoms, co-morbidities, biomarkers of fibrosis and neurohormonal activation. Elevated levels of sST2 are acknowledged as a predictor of worse prognosis in both HF with reduced ejection fraction (HFrEF) and HFpEF. We assume that colchicine decreases inflammation and reduces sST2 levels in HFpEF.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age, male and female
* Left ventricular ejection fraction (LVEF) ≥ 50%
* Symptoms and signs of heart failure
* N-terminal pro-B-type natriuretic peptide (NT-proBNP) ≥300 pg/ml at baseline (patients in atrial fibrillation at baseline NT-proBNP ≥ 600 pg/ml), left atrial volume index (LAVI) >34 mL/m2 or a left ventricular mass index (LVMI) =115 g/m2 for males and =95 g/m2 for females
* body mass index (BMI) > 30kg/m2 or diabetes mellitus

Exclusion Criteria:

* Hypertrophic cardiomyopathy, constrictive pericarditis, or cardiac amyloidosis
* Acute decompensation of HF in the last 1 month
* Valvular heart disease
* Prior history of LVEF below 50%
* Acute myocardial infarction in the last 3 months, cardiac surgery or cerebrovascular accident within the recent 6 months
* Any active or chronic inflammatory diseases or infections
* Patients with indication for colchicine therapy or history of colchicine intolerance
* Severe hepatic (alanine aminotransferase N3 upper limit of normal or renal dysfunction (estimated glomerular filtration rate <45 mL/min per 1.73m2)
* Severe nervous system diseases
* History of any malignancy or suffering from cancer
* Lack of informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Soluble suppression of tumourigenicity 2 (sST2,ng/ml) | from baseline to 12 weeks of treatment
  Delta_circulating sST2

SECONDARY OUTCOMES:
Change in high-sensitivity C-reactive protein (hsCRP, mg/l ) | from baseline to 12 weeks of treatment
  Delta_ circulating hsCRP
Change in N-terminal pro-brain natriuretic peptide (NTproBNP, ng,ml) | from baseline to 12 weeks of treatment
  Delta_circulating NTproBNP
Change in E/e' (average) | from baseline to 12 weeks of treatment
  Delta_ E/e' (average) by 2D- echocardiography
Change in Left ventricular global longitudinal strain (LVGLS,%) | from baseline to 12 weeks of treatment
  Delta_ left ventricular global longitudinal strain by 2D speckle tracking-echocardiography
Left atrial reservoir strain (LA reservoir strain ,%) | from baseline to 12 weeks of treatment
  Delta_ LA reservoir strain by 2D speckle tracking-echocardiography
Drug discontinuation | during 12 weeks of treatment
  Frequency of drug discontinuation
Incidence of side effects | during 12 weeks of treatment
  Side effects will be registered and include gastrointestinal symptoms, hepatotoxicity, muscle weakness or pain, myotoxicity, renal dysfunction
Change in insulin-like growth factor-binding protein 7 (IGFBP-7, ng/ml) | from baseline to 12 weeks of treatment
  Delta_circulating IGFBP-7
Change in procollagen type I carboxy-terminal propeptide (PICP, ng/ml) | from baseline to 12 weeks of treatment
  Delta_circulating PICP
Change in C-terminal telopeptide of collagen type I (CITP,ng/ml) | from baseline to 12 weeks of treatment
  Delta_circulating CITP

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Shchendrygina, Principal Investigator — Sechenov Univerity
Locations (2):
- Russia (2):
  - A Shchendrygina, Moscow
  - Anastasia Shchendrygina, Moscow

REFERENCES:
- [Derived] Shchendrygina A, Rachina S, Cherkasova N, Suvorov A, Komarova I, Mukhina N, Ananicheva N, Gasanova D, Sitnikova V, Koposova A, Smirnova J, Moiseewa E, Drogashevskaya D. Colchicine in patients with heart failure and preserved left ventricular ejection fraction: rationale and design of a prospective, randomised, open-label, crossover clinical trial. Open Heart. 2023 Aug;10(2):e002360. doi: 10.1136/openhrt-2023-002360. PMID 37586845